CLINICAL TRIAL: NCT07303192
Title: The Effect of Injectable Platelet-Rich Fibrin and Low-Level Laser Therapy on Graft Shrinkage in Free Gingival Grafts: A Randomized Controlled Clinical Trial
Brief Title: Effect of i-PRF and LLLT on Free Gingival Graft Shrinkage
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kahramanmaras Sutcu Imam University (Other)
Responsible Party: Principal Investigator, Esra Bozkurt, Assistant Professor, Kahramanmaras Sutcu Imam University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2024/84
Record Dates: First submitted 2025-12-11; First posted 2025-12-24 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Graft Shrinkage; Gingival Recession, Localized
Keywords: free gingival graft; shrinkage; low-level laser therapy; injectable platelet-rich fibrin
MeSH Terms: conditions — Gingival Recession | interventions — proliferation regulatory factors, human urine; Low-Level Light Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control Group (Active Comparator): Patients receive free gingival graft only without additional treatment.
  Interventions: Procedure: Free Gingival Graft (FGG)
- i-PRF group (Experimental): Patients receive free gingival graft with injectable platelet-rich fibrin applied to the graft surface.
  Interventions: Procedure: Free Gingival Graft (FGG); Device: Low-Level Laser Therapy (LLLT)
- LLLT Group (Experimental): Patients receive free gingival graft with low-level laser therapy applied immediately after surgery and on postoperative days 3, 5, 7, and 14.
  Interventions: Procedure: Free Gingival Graft (FGG); Biological: Injectable Platelet-Rich Fibrin (i-PRF)

INTERVENTIONS:
Procedure: Free Gingival Graft (FGG) — Standard free gingival graft procedure performed without additional treatments.
Biological: Injectable Platelet-Rich Fibrin (i-PRF) — Autologous platelet-rich fibrin gel is applied to the graft surface after free gingival graft surgery to potentially reduce graft shrinkage.
  Arms: LLLT Group
Device: Low-Level Laser Therapy (LLLT) — Low-level laser therapy is applied to the graft site immediately after surgery and on postoperative days 3, 5, 7, and 14 to potentially improve healing and reduce graft shrinkage.
  Arms: i-PRF group

SUMMARY:
This randomized clinical trial aims to evaluate whether injectable platelet-rich fibrin (i-PRF) and low-level laser therapy (LLLT) can reduce graft shrinkage after free gingival graft procedures. Free gingival grafts are commonly used to increase the width of keratinized tissue around teeth, but the graft often shrinks during healing. In this study, patients will receive standard free gingival graft surgery with or without additional i-PRF or laser therapy. The goal is to determine whether these treatments improve healing and help maintain the size of the graft.

DETAILED DESCRIPTION:
This randomized controlled clinical trial investigates the effects of injectable platelet-rich fibrin (i-PRF) and low-level laser therapy (LLLT) on the shrinkage of free gingival grafts (FGG) used to treat gingival recession. Free gingival grafting is commonly performed to increase the width of keratinized tissue around teeth, but shrinkage during healing can reduce clinical outcomes.

The study included 48 systemically healthy adult patients with Cairo Class I gingival recession in mandibular anterior teeth. Participants were randomly assigned to one of three groups: control (FGG alone), i-PRF (FGG + platelet-rich fibrin), or LLLT (FGG + low-level laser therapy). Ethical approval was obtained from the Clinical Research Ethics Committee of Inonu University (Protocol No: 2024/84), and all participants provided written informed consent. The study protocol was registered at ClinicalTrials.gov (NCT06744270) and conducted according to CONSORT 2010 guidelines.

All patients received preoperative periodontal treatment, including plaque removal and oral hygiene instructions. Free gingival grafts were harvested from the palatal region and adapted to the recipient site, then stabilized with sutures. In the i-PRF group, autologous platelet-rich fibrin gel was applied to the graft surface. In the LLLT group, laser therapy was applied immediately after surgery and on postoperative days 3, 5, 7, and 14. The control group received no additional treatment beyond standard grafting.

Postoperative care included use of a periodontal dressing, chlorhexidine mouthwash, analgesics as needed, and oral hygiene instructions after suture removal. Clinical evaluations included gingival recession depth, keratinized tissue height, probing depth, clinical attachment level, and graft area measurements at baseline, 1, 3, and 6 months. Edema, erythema, and patient-reported pain were also assessed during follow-up.

The primary outcome of the study was graft shrinkage, calculated as the percentage decrease in graft area over time. Secondary outcomes included clinical parameters and patient-reported postoperative morbidity. All measurements were performed by calibrated, blinded examiners to ensure reliability.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years.
* Systemically healthy.
* Cairo Class I gingival recession in vital mandibular anterior incisors.
* No caries or restorations in the relevant teeth.
* Keratinized gingiva height < 2 mm in the included teeth.
* Plaque Index (PI) < 1.
* Gingival Index (GI) < 1.

Exclusion Criteria:

* Active periodontal disease or probing depth > 3 mm.
* Use of medications that could prevent surgery or affect wound healing.
* Pregnancy or breastfeeding.
* History of periodontal surgery in the working area.
* Active smokers.
* Current orthodontic treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2024-07-01 (Actual); Primary Completion 2025-08-30 (Actual); Study Completion 2025-08-30 (Actual)

PRIMARY OUTCOMES:
Graft Area Shrinkage (%) | Baseline, 1 month, 3 months, and 6 months postoperatively.
  Change in graft surface area, expressed as percentage shrinkage from baseline. Standardized clinical photographs taken at baseline and at postoperative 1, 3, and 6 months were analyzed using calibrated digital image analysis software (ImageJ). The graft borders were traced, and surface area (mm²) was calculated. Each measurement was repeated three times, and the mean value was used. Shrinkage percentage was calculated using the formula:
  Shrinkage % = [(baseline area - follow-up area) / baseline area] × 100.
Root Coverage Percentage (%) | Baseline and 6 months postoperatively.
  Percentage of root coverage obtained at 6 months. Root coverage was calculated from changes in gingival recession depth (RD) using the formula:
  Root Coverage % = [(baseline RD - RD at 6 months) / baseline RD] × 100. RD was defined as the distance from the CEJ to the gingival margin and measured using a manual periodontal probe.
Gingival Recession Depth (RD) | Baseline, 1 month, 3 months, and 6 months postoperatively.
  Change in gingival recession depth measured in millimeters.
Keratinized Tissue Height (KTH) | Baseline, 1 month, 3 months, and 6 months postoperatively.
  Change in keratinized tissue height measured in millimeters.

SECONDARY OUTCOMES:
Probing Depth (PD) | Baseline, 1 month, 3 months, and 6 months postoperatively.
  Change in probing depth measured in millimeters.
Clinical Attachment Level (CAL) | Baseline, 1 month, 3 months, and 6 months postoperatively.
  Change in clinical attachment level measured in millimeters.
Oedema Score in the Recipient Site | Postoperative days 3, 5, 7, 14, 21, and 28.
  Oedema was scored clinically in the recipient area using a 0-4 ordinal scale (0 = none; 1 = mild, intraoral oedema limited to the surgical site; 2 = moderate, extraoral oedema limited to the surgical site; 3 = significant, extraoral oedema extending beyond the surgical site; 4 = severe, extraoral oedema extending beyond the surgical site with limited mouth opening). Examinations were performed by a calibrated and blinded examiner. Higher scores indicate more severe oedema.
  Unit of Measure: Units on a scale (0-4)
Erythema Score in the Recipient Site | Postoperative days 3, 5, 7, 14, 21, and 28.
  Erythema was scored clinically in the recipient area using a 0-4 ordinal scale (0 = none, tissues fully pink; 1 = mild, <25% of tissues red; 2 = moderate, 25-50% of tissues red; 3 = significant, 50-75% of tissues red; 4 = severe, >75% of tissues red). Examinations were performed by a calibrated and blinded examiner. Higher scores indicate greater severity of erythema.
Pain Intensity (VAS Score) | First postoperative week.
  Postoperative pain intensity was assessed using a 0-10 Visual Analog Scale (VAS), where 0 = no pain and 10 = maximum tolerable pain. Patients recorded their pain level daily during the first postoperative week. Higher scores indicate greater pain intensity.
Analgesic Consumption | First postoperative week.
  The number of analgesic tablets taken during the first postoperative week was recorded by each patient on a provided daily log form. Higher values indicate greater postoperative analgesic use.

CONTACTS AND LOCATIONS:
Overall Officials: esra bozkurt, Principal Investigator — Kahramanmaras Sutcu Imam University
Locations (1):
- Kahramanmaraş Sütçü İmam University, Kahramanmaraş, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared to ensure patient privacy and confidentiality.

REFERENCES:
- [Background] Shakiliyeva S, Sahin D, Gunpinar S, Gursel M. Comparison of conventional and modified sling suture techniques in free gingival graft operations-a randomized controlled clinical trial. BMC Oral Health. 2025 Feb 21;25(1):279. doi: 10.1186/s12903-025-05456-x. PMID 39984903
- See also: Inonu University Clinical Research Ethics Committee — https://www.inonu.edu.tr/klinik.etik